CLINICAL TRIAL: NCT03853343
Title: Pilot Exploratory Investigation Into the Effects of Brown Seaweed Extract Supplementation on Metabolic Biomarkers
Brief Title: Seaweed Extract Supplementation and Metabolic Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioAtlantis Ltd. (Industry)
Collaborators: University of Roehampton (Other)
Responsible Party: Principal Investigator, Dr. George Tzortzis, Principle Investigator Human Health, BioAtlantis Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BioAtlDG001
Record Dates: First submitted 2019-01-22; First posted 2019-02-25 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome; Insulin Sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 3 capsules per day (1 before each meal) of cellulose
  Interventions: Dietary Supplement: Placebo
- Seaweed extract (Active Comparator): 3 capsules per day (1 before each meal) of seaweed extract
  Interventions: Dietary Supplement: Seaweed extract

INTERVENTIONS:
Dietary Supplement: Seaweed extract — 1 capsule 3 times per day
  Arms: Seaweed extract
Dietary Supplement: Placebo — 1 capsule 3 times per day
  Arms: Placebo

SUMMARY:
Double blinded, randomized, placebo controlled preliminary pilot exploratory investigation into the effects of brown seaweed extract supplementation, on fasting blood Insulin, fasting blood glucose, insulin sensitivity, blood inflammatory markers and tolerance in healthy overweight adults.

DETAILED DESCRIPTION:
Diabetes melitus is a group of metabolic disorders resulting from a defect in insulin production and/or insulin action. The World Health Organisation (WHO) has estimated that the total number of people with diabetes mellitus worldwide will increase from 171 million in 2000 to nearly 370 million in 2030 with the prevalence of the disease for all age groups to be 4.4%. 90% of diabetes cases worldwide are of Type II diabetes mellitus (T2DM) as a result of greater prevalence of sedentary lifestyle, unhealthy diet and rise of obesity, as well as an increasing number of elderly population. T2DM can be attributed to relative deficiency of insulin, involving insulin resistance, aberrant synthesis of hepatic glucose and progressive deterioration of pancreatic beta-cell functions resulting in chronic hyperglycaemia with disturbances in carbohydrate, fat and protein metabolism. Insulin resistance, classically defined as a decreased sensitivity to metabolic actions of insulin, is recognised as an important risk factor in the pathogenesis of various disorders, including T2DM. However, insulin resistance and ß-cell dysfunction can be asymptomatic and may remain undiagnosed for many years. Current T2DM management employs a range of pharmacological (hypoglycaemic agents) and lifestyle (diet, exercise) intervention approaches aiming at managing hyperglycaemia, with the main objective being to ensure sufficient delivery of glucose to the various tissues of the body and prevent hyperglycaemia by achieving good glycemic control. Nutrition has been regarded to play a significant role in the complex pathophysiology of T2DM and in the last several years, increasing amount of evidence has emerged linking various nutrients and food sources with a positive management of T2DM.

Seaweed have traditionally been consumed as a readily available whole food or traditional medical preparations, especially in Asia. Seaweeds are rich in bioactive compounds in the form of polyphenols, carotenoids, vitamins, minerals, phycobilins, phycocyanins, and polysaccharides, many of which are known to offer a wide range of benefits in human health.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 25-35 kg/m2
* Not dieting within the last month and not having lost >5% body weight in the previous year
* Not increased physical activity levels in the past 2-4 weeks or intending to modify them during the study
* Understands and is willing, able and likely to comply with all study procedures and restriction including being willing to follow the nutritional advice
* Able to eat most everyday foods
* Habitually consumes three standard meals a day

Exclusion Criteria:

* Significant health problems (e.g. hypercholesterolaemia, diabetes, GI disorders)
* Taking any medication or supplements known to affect mineral or glucose metabolism within the past month and/or during the study
* Pregnant, planning to become pregnant or breastfeeding
* History of anaphylaxis to food
* Known allergies or intolerance to foods and/or to the study materials (or closely related compounds) or any of their stated ingredients
* BMI <25 kg/m2 or >35 kg/m2
* Volunteers self-reporting currently dieting or having lost >5% body weight in the previous year
* Participants with abnormal eating behaviour
* Participation in another experimental study or receipt of an investigational drug/product within 30 days of the screening visit
* Volunteers who have significantly changed their physical activity in the past 2-4 weeks or who intend to change them during the study
* Participants receiving systemic or local treatment likely to interfere with the evaluation of the study parameters
* Participants on specific food avoidance diets
* Participants who work in appetite or feeding related areas

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Glucose concentration | 3 weeks
  Changes in plasma glucose in healthy volunteers with BMI>25 after 3 weeks of treatment
Change of Plasma Insulin concentration | 3 weeks
  Changes in plasma insulin in healthy volunteers with BMI>25 after 3 weeks of treatment
Change in metabolic parameters | 3 weeks
  Changes in insulin sensitivity based on Homeostasis Model Assessment- Insulin Resistance (HOMA-IR) test

SECONDARY OUTCOMES:
Change in Blood Lipids | 3 weeks
  Changes in total cholesterol, HDL-C and triglycerides following 3 weeks supplementation
Change in plasma Markers of inflammation | 3 weeks
  Changes in Tumor Necrosis Factor-alpha, Interleukin-6, Interleukin-1b, Interleukin-10, Interferon-gamma and C-Reactive Protein following 3 weeks of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: George Tzortzis, Study Director — BioAtlantis Ltd.
Locations (1):
- Roehampton University, London, United Kingdom